CLINICAL TRIAL: NCT05548166
Title: Phase 1 Protocol to Develop a Patient-reported Outcome Measure for Children and Adolescents With Celiac Disease: CELIAC-Q KIDS
Brief Title: Development of CELIAC-Q KIDS: A Patient-Reported Outcome Measure for Pediatric Celiac Disease
Status: Active, not recruiting | Type: Observational
Sponsor: McMaster University (Other)
Collaborators: The Hospital for Sick Children (Other); Canadian Celiac Association (Unknown)
Responsible Party: Sponsor
Other Study IDs: 11126
Record Dates: First submitted 2022-09-16; First posted 2022-09-21 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Celiac Disease in Children; Celiac Disease; Patient-reported Outcome Measures
MeSH Terms: conditions — Celiac Disease | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Pediatric Patients: Pediatric patients with celiac disease.
  Interventions: Other: Interview and scale development
- Caregivers and parents: Caregivers and parents of pediatric patients with celiac disease
  Interventions: Other: Interview and scale development
- Experts: Group of experts in pediatric celiac disease to provide feedback on scale development.
  Interventions: Other: Interview and scale development

INTERVENTIONS:
Other: Interview and scale development — Interview and scale development

SUMMARY:
A multicentre, prospective observational study to develop the CELIAC-Q KIDS patient reported outcome measure for children and adolescents with celiac disease. The CELIAC- Q KIDS will contain a comprehensive set of independently functioning scales designed to measure outcomes that matter to children with celiac disease, as well as scales to measure patients experience with the gluten-free diet.

DETAILED DESCRIPTION:
The study will be conducted in three stages:

Stage I - Conceptual framework development: A scoping review will be carried out to map initial concepts that have been measured by patient report in pediatric patients with celiac disease. Findings will be used to develop a preliminary conceptual framework.

Stage II - Item generation: Approximately 20 interviews will be conducted with children and adolescents with celiac disease and their caregivers to capture their experiences including quality of life, symptom experience, and other relevant themes that may emerge. The interviews will be audio recorded and transcribed verbatim. The qualitative data will be analyzed thematically, and key quotes extracted which will be used to create a draft item list. Interviews will be conducted either in person or virtually depending on patient preference. The data from Stage I will be used to develop a preliminary version of the CELIAC-Q KIDS patient-reported outcome measure.

Stage II - Scale refinement:

The CELIAC-Q KIDS scales will be refined through multiple rounds of cognitive debriefing interviews using the "think aloud method." During each interview round, approximately 7 children and adolescents with celiac disease will be interviewed to determine if patients understand the instructions, response options and items of the CELIAC-Q KIDS instrument and to identify missing content. Interviews will take place in a series of rounds to allow time to make changes to the instrument and then obtain feedback on those changes until data saturation is achieved.

Between rounds of cognitive debriefing interviews, the CELIAC-Q KIDS will be shown to experts for feedback. A multidisciplinary, international group of approximately 10 healthcare providers who care for children and adolescents with celiac disease will be surveyed to determine if healthcare providers feel there are any items missing from the patient-reported outcome measure, if any items are not relevant and to provide feedback on the instructions and response options. Once again, feedback provided by the experts will be used to revise the CELIAC-Q KIDS scales.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with celiac disease.
* Pediatric patients (18 years and younger).
* Ability to understand and communicate in the English language

Exclusion Criteria:

* Patients who do not have celiac disease.
* Non-pediatric patients (over 18).
* Unable to understand and communicate in the English language

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — Patients of all genders are included in this study.
Study Population: This study will include participants from the McMaster Children's Hospital Pediatric Celiac Disease Clinic and the Hospital for Sick Children (SickKids) Children's Celiac Clinic. Patients who have confirmed celiac disease (based on biopsy and/or serology) will be recruited to participant. Patients aged 1 to 8 years of age will participate in the interviews with their caregiver, whereas caregivers will participate on their own when their child is under the age of 8. Both genders will be recruited in patient and parent groups.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-10-26 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Development of the patient-reported outcome measure: Consensus on items that will comprise the newly developed disease-specific patient-reported outcome measure for pediatric celiac disease | 48 Months
  Development of the CELIAC-Q KIDS scales: qualitative interview and survey-based data will be analyzed qualitatively to develop and refine the items that comprise the scales

SECONDARY OUTCOMES:
Qualitative interviews - for item generation | 24 months
  Patient participants
Cognitive debriefing interviews - qualitative feedback on scale instructions, response options and items | 24 months
  Patient participants
Expert survey data - qualitative feedback on scale instructions, response options and items | 24 months
  Expert participant questionnaire

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - McMaster Children's Hospital, Hamilton, Ontario
  - SickKids | The Hospital for Sick Children, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Undecided